CLINICAL TRIAL: NCT02104232
Title: Thinking Healthy Program - Peer Delivered, India (THPP-I)
Acronym: THPP-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THPP-I MH095687; 1U19MH095687-01 (NIH)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Unipolar Depression
Keywords: Maternal depression
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THPP-I (Experimental): TPs in the THPP-I group receive, in addition to enhanced usual care (EUC), between 6 to 14 sessions of THPP (simple cognitive behaviour therapy) starting from their recruitment in the second/ third trimester until up to 6 months after child birth. Sessions will be delivered by peers on an individual basis at a location of convenience to the TPs.
  Interventions: Behavioral: THPP-I; Behavioral: EUC
- Enhanced usual care (EUC) (Other): Enhanced usual care (EUC) will comprise communicating the results of the screening to the mother through an information sheet on self-care for mental health, communicating the results to the mother's gynaecologist, providing the gynaecologist with the WHO mental health gap (mhGAP) guidelines for the treatment of depression, and providing guidance on referral of depressed mothers to mental health services.
  Interventions: Behavioral: EUC

INTERVENTIONS:
Behavioral: THPP-I
  Arms: THPP-I
Behavioral: EUC

SUMMARY:
Background The rates of perinatal depression in South Asian women are reported to be amongst the highest in the world, ranging from 18%-30% in urban areas and 28%-36% in rural areas. In addition to its profound impact on women's health, disability and functioning, perinatal depression is associated with poor child health outcomes such as pre-term birth, infant under-nutrition and stunting. There is robust evidence that perinatal depression can be effectively managed with psychological treatments delivered by non-specialist health care workers. The Thinking Healthy Program (THP), a psychological treatment delivered by community health workers (CHWs) in Pakistan, more than halved the rate of perinatal depression among mothers and led to significant improvements in child health outcomes. To enhance access to such evidence-based psychological treatments there is a need to examine the potential role of other human resources such as lay persons in delivering psychological treatments such as THP in poor resource settings.

Objective To evaluate the effectiveness and cost-effectiveness of THP delivered by peers (the Thinking Healthy Program-Peer delivered in Goa, India; THPP-I) over the duration of 6 months. Peers will be healthy mothers who live in the same community as potential trial participants (TPs).

Study design and outcomes Individual randomized controlled trial in Goa, India involving 280 women. TPs will not be blinded to treatment allocation. Mothers attending antenatal clinics at hospitals will be assessed for eligibility to participate in the trial (e.g. whether they are in the second or third trimester of pregnancy). Those who are eligible will be invited to participate in screening for depression; mothers who consent will be screened for depression with a locally validated version of the Patient Health Questionnaire (PHQ-9). Women who screen positive (PHQ-9 score ≥ 10) and give informed consent for further participation in the trial will be randomly allocated in a 1:1 ratio to receive enhanced usual care (EUC) or THPP-I+EUC, using a computer generated allocation sequence. The primary outcomes will be remission (i.e. recovery from depression and depressive symptoms), both assessed by the PHQ-9 at 6 months. Secondary outcomes are depressive symptoms and remission at 3 months (PHQ-9), maternal disability at 3 and 6 months (measured with the WHO-DAS), perceived social support, breastfeeding rates and infant weight and height of children at 3 and 6 months. Outcomes will be analyzed on an intention to treat basis.

Interventions EUC will comprise communicating the results of the screening to the mother through an information sheet on self-care for mental health, communicating the results to the mother's gynaecologist, providing the gynaecologist with the WHO mhGAP guidelines for the treatment of depression, and providing guidance on referral of depressed mothers to mental health services. TPs who are in the THPP-I group will receive, in addition to EUC, between 6 to 14 sessions of THPP starting from their recruitment in the second/ third trimester until up to 6 months after child birth. Sessions will be delivered by peers on an individual basis at a location of convenience to the TPs (usually at their own homes).

Implications THPP-I has the potential to advance knowledge of the extent to which task-shifting of the delivery of evidence-based psychological treatments can be extended to peers in the community. If effectiveness is observed, this approach offers a potential opportunity to access a vast untapped human resource for maternal mental health care and addresses a major barrier in global mental health - the lack of skilled and motivated human resources in the formal health sector - offering a new avenue for the scaling up of evidence-based psychological treatments and mental health services in low resourced settings.

ELIGIBILITY:
Inclusion Criteria:

* In the 2nd or 3rd trimester of pregnancy
* Aged 18 years and over
* Intending to reside in the selected areas of the intervention delivery for the entire duration of the study (mothers intending to be away for more than 2 months during or after the period of child birth will be excluded).

Exclusion criteria:

* Mothers requiring immediate inpatient care for any reason (medical or psychiatric)
* Mothers who do not speak any of the following languages: Konkani, Hindi, English, Marathi
* Mothers whose expected date of delivery is within 3 weeks of their screening date
* Previously screened using the PHQ-9 within the last month
* Mothers with difficulty hearing/speaking which makes the assessment difficult

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Remission (i.e. recovery from depression) and depressive symptoms, assessed by the PHQ-9 | 6 months post-child birth

SECONDARY OUTCOMES:
Depressive symptoms and remission (PHQ-9) | 3 months post-child birth
Maternal disability (measured with the WHO-DAS) | 3 and 6 months post-child birth
Breastfeeding rates of women | 3 and 6 months post child birth
Infant weight | 3 and 6 months post-child birth
Infant height | 3 and 6 months post child birth
Perceived social support (measured with MSPSS) | 3 and 6 months post child birth

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Sangath, Goa, India

REFERENCES:
- [Derived] Vanobberghen F, Weiss HA, Fuhr DC, Sikander S, Afonso E, Ahmad I, Atif N, Bibi A, Bibi T, Bilal S, De Sa A, D'Souza E, Joshi A, Korgaonkar P, Krishna R, Lazarus A, Liaqat R, Sharif M, Weobong B, Zaidi A, Zuliqar S, Patel V, Rahman A. Effectiveness of the Thinking Healthy Programme for perinatal depression delivered through peers: Pooled analysis of two randomized controlled trials in India and Pakistan. J Affect Disord. 2020 Mar 15;265:660-668. doi: 10.1016/j.jad.2019.11.110. Epub 2019 Nov 23. PMID 32090783
- [Derived] Fuhr DC, Weobong B, Lazarus A, Vanobberghen F, Weiss HA, Singla DR, Tabana H, Afonso E, De Sa A, D'Souza E, Joshi A, Korgaonkar P, Krishna R, Price LN, Rahman A, Patel V. Delivering the Thinking Healthy Programme for perinatal depression through peers: an individually randomised controlled trial in India. Lancet Psychiatry. 2019 Feb;6(2):115-127. doi: 10.1016/S2215-0366(18)30466-8. PMID 30686385
- [Derived] Atif N, Krishna RN, Sikander S, Lazarus A, Nisar A, Ahmad I, Raman R, Fuhr DC, Patel V, Rahman A. Mother-to-mother therapy in India and Pakistan: adaptation and feasibility evaluation of the peer-delivered Thinking Healthy Programme. BMC Psychiatry. 2017 Feb 23;17(1):79. doi: 10.1186/s12888-017-1244-z. PMID 28231791
- [Derived] Sikander S, Lazarus A, Bangash O, Fuhr DC, Weobong B, Krishna RN, Ahmad I, Weiss HA, Price L, Rahman A, Patel V. The effectiveness and cost-effectiveness of the peer-delivered Thinking Healthy Programme for perinatal depression in Pakistan and India: the SHARE study protocol for randomised controlled trials. Trials. 2015 Nov 25;16:534. doi: 10.1186/s13063-015-1063-9. PMID 26604001